CLINICAL TRIAL: NCT05416164
Title: DESCARTES: De-ESCAlation of RadioTherapy in Patients With Pathologic Complete rESponse to Neoadjuvant Systemic Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other); Borstkanker Onderzoek Groep (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21CAR
Record Dates: First submitted 2022-04-19; First posted 2022-06-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant Chemotherapy; Breast cancer; Complete response; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omission of radiotherapy (Experimental)
  Interventions: Radiation: Omission of radiotherapy

INTERVENTIONS:
Radiation: Omission of radiotherapy — Omission of radiotherapy

SUMMARY:
This study evaluates whether radiotherapy can safely be omitted in breast cancer patients with T1-2N0 tumors who achieve a pathologic complete response after neoadjuvant systemic therapy and breast-conserving surgery

DETAILED DESCRIPTION:
The proportion of women diagnosed with breast cancer who are treated with neoadjuvant systemic therapy is increasing. Depending on the subtype, 10-75% of these patients will have a pathologic complete response. Currently breast conserving surgery with pathologic complete response is followed by radiotherapy. In this patient group risk of local recurrence is low, but radiotherapy may cause considerable morbidity.

The aim of this study is to investigate whether omitting radiotherapy is safe for patients with a node-negative breast tumor <5cm treated with neoadjuvant systemic therapy and breast conserving surgery who achieve a pathologic complete response

ELIGIBILITY:
Inclusion Criteria:

* Women, aged ≥ 18 years
* Invasive HR positive/Her2 negative, Her2+ (ER/PR +/-) or TN breast cancer
* Concurrent DCIS in pre-NST biopsy is allowed if there is no suspicion of extensive component i.e. absence of non-mass enhancement on pre-NST MRI, contrast-enhanced mammography or breast-specific gamma imaging and/or absence of calcifications on pre-NST mammography
* Primary tumour (T) clinical stage cT1-2
* Unifocal disease; confirmed by pre-NST MRI, contrast-enhanced mammography or breast-specific gamma imaging
* Clinical nodal stage 0; absence of lymph node metastases should be confirmed by ultrasound or FDG-PET/CT
* Neoadjuvant systemic treatment (NST)
* Marker placed in breast tumour prior to NST
* Breast conserving surgery performed, i.e. no mastectomy
* Sentinel node biopsy performed before or after NST
* Pathologic complete response in breast and lymph nodes, i.e. no residual tumour cells or DCIS detected
* Written informed consent

Exclusion Criteria:

* Primary tumour (T) clinical stage cT3-4
* Pre- or post-NST diagnosis of nodal disease including isolated tumour cells
* Patients without axillary ultrasound or FDG-PET/CT pre-NST
* History of breast cancer or DCIS
* Synchronous contralateral breast cancer or DCIS
* Synchronous M1 disease
* Carrier of gene mutation associated with increased risk of breast cancer, i.e. BRCA1, BRCA2, CHEK2, TP53 or PALB-2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2037-05 (Estimated)

PRIMARY OUTCOMES:
Local recurrence | 5 years
  To show that radiotherapy after neoadjuvant systemic therapy and breast-conserving surgery can be omitted in T1-2N0 breast cancer patients who achieve pathologic complete response without compromising the 5 - year local recurrence rate (i.e, < 6% axillary recurrences within 5 years).

SECONDARY OUTCOMES:
Level of cancer worry | 4 years
  The patients' experienced level of cancer worry will be measured using the validated 8-item Cancer Worry Scale (i.e., low (Cancer Worry Scale score ≤ 13 at each assessment) and high (Cancer Worry Scale score ≥14 at each assessment)).
Satisfaction reported by PROM (patient reported outcome measures) | 4 years
  The patients´experienced quality of life and satisfaction will be measured using the validated questionnaire EORTC-QLQ-C30 (Quality of life in cancer patients) and EORTC-QLQ-BR23 (Quality of life of patients with breast cancer)
Overall survival | 5 and 10 years
Disease-specific survival | 5 and 10 years
Locoregional recurrence | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Hemert AKE, van Olmen JP, Boersma LJ, Maduro JH, Russell NS, Tol J, Engelhardt EG, Rutgers EJT, Vrancken Peeters MTFD, van Duijnhoven FH. De-ESCAlating RadioTherapy in breast cancer patients with pathologic complete response to neoadjuvant systemic therapy: DESCARTES study. Breast Cancer Res Treat. 2023 May;199(1):81-89. doi: 10.1007/s10549-023-06899-y. Epub 2023 Mar 9. PMID 36892723

DOCUMENTS (1):
  • Study Protocol (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT05416164/Prot_000.pdf